CLINICAL TRIAL: NCT03578016
Title: A Randomized and Controlled Trial Using Circle of Security-Parenting for Parents of Children Referred to Child Psychiatric Services.
Brief Title: COS-P for Parents of Children Referred to Child Psychiatric Services
Acronym: COS-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Syddanmark (Other)
Responsible Party: Principal Investigator, Aida Bikic, assistant professor, ph.d., Region Syddanmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-58-0035
Record Dates: First submitted 2018-04-08; First posted 2018-07-05 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Child Behavior Problem
Keywords: attachment; parent; training; sensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circle of Security-Parenting (Experimental): 10 weekly, manualized group sessions at the clinic
  Interventions: Other: Circle of Security-Parenting; Other: Treatment as Usual
- Treatment as Usual (TAU) (Other): TAU consists of clinical assessment and treatment.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Circle of Security-Parenting — COS-P is a brief, behavioral and insight oriented therapeutic group approach for parents with the aim to promote parental sensitivity and attachment and autonomy in the parent-child relationship. The parents will participate in ten weekly 1,5-hour sessions at the clinic conducted by two COS-certified therapists. Groups will include 4-5 families at a time.
  Other Names: COS-P
  Arms: Circle of Security-Parenting
Other: Treatment as Usual — TAU consists of clinical assessment and treatment.
  Other Names: TAU

SUMMARY:
Background:The quality of attachment is greatly influenced by parental sensitivity. Attachment based interventions are designed to promote parental sensitivity, to change parental mental representations and to improve understanding of the developmental needs of the child. Very few studies have investigated the effect of attachment-based interventions on psychiatric symptoms in children. Targeting parental sensitivity and the parent-child interaction might have an important impact on psychiatric symptoms in a clinical sample of children referred to child psychiatric services.

Objectives: The primary objective is to investigate whether Circle of Security-Parenting (COS-P) has an effect on parental sensitivity in parents of children referred to child psychiatric services. The secondary objectives are to investigate the effect on children's behavioral and emotional symptoms and the parental stress and reflective functioning after 10 weeks of intervention and at the 24 week follow-up. The study is also exploring the effect of parental attachment style, parental stress and parental psychopathology on the effect of the intervention.

Methods: The trial will include 128 families of children (age 3-8 years) who are referred to child psychiatric services in a randomized and controlled design. Included families will be randomized to COS-P+ Treatment as Usual (TAU) or TAU only.

Perspectives: Considering the important impact of the quality of the parent-child relationship on the child's well-being, it is essential to target it in interventions and to investigate the relation with psychiatric symptoms. Generally there is a lack of interventions targeting parental sensitivity in psychiatric child populations. Working with the parents on the child-parent relation, might have an important impact on their children's current psychiatric symptoms and could additionally prevent future psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* Children who score equal or above the 93d percentile on CBCL-total score
* Score above 93d percentile on the CBCL- ODD or aggression scale
* Informed consent from both custody.

Exclusion Criteria:

For children:

* autism spectrum disorders
* serious psychopathology requiring immediate clinical attention
* head injury or verified neurological disease
* intelligence quotient (IQ) <80
* medical condition, requiring treatment
* no informed consent from custody

For parents:

* a diagnosis of schizophrenia
* bipolar disorder
* known substance abuse
* severe intellectual impairment
* suicide attempt in the past

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Maternal sensitivity | after 10 weeks of intervention
  Maternal sensitivity is measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)

SECONDARY OUTCOMES:
Maternal Intrusiveness | after 10 weeks of intervention
  Measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)
Maternal Sensitivity | 24 week follow-up
  Measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)
Maternal Intrusiveness | 24 week follow-up
  Measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)
Dyadic reciprocity | after 10 weeks of intervention
  Measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)
Dyadic reciprocity | 24 week follow-up
  Measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)
Negative states | after 10 weeks of intervention
  Measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)
Negative states | 24 week follow-up
  Measured by observing a mother-child interaction and is rated using "Coding Interactive Behavior" (CIB)
Child Behaviour Check List (CBCL)-Total score-parent rated | after 10 weeks of intervention
  Parent questionnaire on child symptoms. Score range (0-236). Higher indicates more problems.
Child Behaviour Check List (CBCL)-Total score-parent rated | 24 week follow-up
  Parent questionnaire on child symptoms. Score range: 0-236. Higher indicates more problems.
CBCL-ODD score-parent rated. Score range: 0-26. Higher indicates more problems. | after 10 weeks of intervention
  Parent questionnaire on child symptoms
CBCL-ODD score-parent rated. Score range: 0-26. Higher indicates more problems. | 24 week follow-up
  Parent questionnaire on child symptoms
Berkeley Puppet interview | after 10 weeks of intervention
  Child interview
Berkeley Puppet interview | 24 week follow-up
  Child interview
Coping with childrens negative emotions scale | baseline
  Parent questionnaire on their strategies coping with children's negative emotions. Score range 72-504.
Coping with childrens negative emotions scale | after 10 weeks of intervention
  Parent questionnaire on their strategies coping with children's negative emotions. Score range 72-504.
Coping with childrens negative emotions scale | 24 week follow-up
  Parent questionnaire on their strategies coping with children's negative emotions. Score range 72-504.
Parental Reflective Functioning Questionnaire | baseline
  Parent self-report measure that assesses parental reflective functioning or mentalizing. Score range 1-126.
Parental Reflective Functioning Questionnaire | after 10 weeks of intervention
  Parent self-report measure that assesses parental reflective functioning or mentalizing. Score range 1-126.
Parental Reflective Functioning Questionnaire | 24 week follow-up
  Parent self-report measure that assesses parental reflective functioning or mentalizing. Score range 1-126.
Eyberg Child Behaviour Inventory (ECBI) | after 10 weeks of intervention
  Parent questionnaire on child behavior. Score range 36-252. Higher indicating more problems.
Eyberg Child Behaviour Inventory (ECBI) | 24 week follow-up
  Parent questionnaire on child behavior. Score range 36-252. Higher indicating more problems.

OTHER OUTCOMES:
Major Depression Inventory- mother and partner | baseline
  Parent questionnaire on their own depressive symptoms. Score range 0-50. Higher scores indicating more severe symptoms.
Revised Adult Attachment Scale (RAAS) | baseline
  Questionnaire regarding the attachment style of the mother and partner. Scofre range 18-90.
Standardized Assessment of Personality (SAPAS)-mother and partner | baseline
  A short and simple interview-administered screen for personality disorders. Score range 1-8, higher score indicating more problems.
Strength and Difficulties Questionnaire (SDQ) | baseline
  Parent questionnaire on the strength and difficulties of the child. Total difficulties score 0-40. Higher indicating more problems.
Strength and Difficulties Questionnaire (SDQ) | after 10 weeks of intervention
  Parent questionnaire on the strength and difficulties of the child. Total difficulties score 0-40. Higher indicating more problems.
Strength and Difficulties Questionnaire (SDQ) | 24 week follow-up
  Parent questionnaire on the strength and difficulties of the child. Total difficulties score 0-40. Higher indicating more problems.
Brief Symptom Inventory | baseline
  Parent questionnaire on their own symptoms. Score range 0-212. Higher indicating more problems.
Attention Deficit Hyperactivity Disorder- Rating Scale (ADHD-RS) | after 10 weeks of intervention
  Parent questionnaire on child ADHD symptoms. Score range: 1-78. Higher indicates more problems.
Attention Deficit Hyperactivity Disorder- Rating Scale (ADHD-RS) | 24 weeks follow up
  Parent questionnaire on child ADHD symptoms. Score range: 1-78. Higher indicates more problems.
Parental Stress Scale | after 10 weeks of intervention
  Parent rating scale on their stress level. Score range: 18-90. Higher scores indicate more stress.
Parental Stress Scale | 24 week follow up
  Parent rating scale on their stress level. Score range: 18-90. Higher scores indicate more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Aida Bikic, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Department of Child and Adolescent Mental Health Services, Aabenraa, Denmark

REFERENCES:
- [Derived] Bikic A, Smith-Nielsen J, Dalsgaard S, Swain J, Fonagy P, Leckman JF. Protocol for a randomized controlled trial comparing the Circle of Security-parenting (COS-P) with treatment as usual in child mental health services. PLoS One. 2022 Apr 26;17(4):e0265676. doi: 10.1371/journal.pone.0265676. eCollection 2022. PMID 35472058